CLINICAL TRIAL: NCT02372370
Title: Pretreatments of the Skin to Enhance MAL-induced Protoporphyrin IX (PpIX) Accumulation Prior to Photodynamic Therapy (PDT)
Brief Title: Pretreatments of the Skin Prior to PDT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Merete Haedersdal, Professor, DMSci, MD, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2014-132
Record Dates: First submitted 2015-02-10; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interventions (Active Comparator): All participants receive all interventions.
  Interventions: Procedure: Microneedle pretreatment + MAL-PDT; Procedure: Sandpaper pretreatment + MAL-PDT; Procedure: Curettage pretreatment + MAL-PDT; Procedure: Ablative Fractional Laser (AFXL) pretreatment + MAL-PDT; Procedure: Non-Ablative Fractional Laser (NAFXL) pretreatment + MAL-PDT; Drug: MAL Control.; Other: Untreated Control

INTERVENTIONS:
Procedure: Microneedle pretreatment + MAL-PDT — Interventions: microneedling of the skin using dermarollers prior to topical application of 125 microliter methyl aminolevulinate (MAL) cream followed by red light illumination after 3 hours incubation (i.e. photodynamic therapy (PDT)). Three settings are applied: mild, moderate and strong.
Procedure: Sandpaper pretreatment + MAL-PDT — Interventions: abrasion of the skin using Abrasive Pads for Skin Preparation prior to topical application of 125 microliter methyl aminolevulinate (MAL) cream followed by red light illumination after 3 hours incubation (i.e. photodynamic therapy (PDT)). Three settings are applied: mild, moderate and strong.
Procedure: Curettage pretreatment + MAL-PDT — Interventions: curettage of the skin using a curette prior to topical application of 125 microliter methyl aminolevulinate (MAL) cream followed by red light illumination after 3 hours incubation (i.e. photodynamic therapy (PDT)). Three settings are applied: mild, moderate and strong.
Procedure: Ablative Fractional Laser (AFXL) pretreatment + MAL-PDT — Interventions: Ablative Fractional Laser (AFXL) resurfacing of the skin prior to topical application of 125 microliter methyl aminolevulinate (MAL) cream followed by red light illumination after 3 hours incubation (i.e. photodynamic therapy (PDT)). Three settings are applied: mild, moderate and strong.
Procedure: Non-Ablative Fractional Laser (NAFXL) pretreatment + MAL-PDT — Interventions: Non-Ablative Fractional Laser (NAFXL) resurfacing of the skin prior to topical application of 125 microliter methyl aminolevulinate (MAL) cream followed by red light illumination after 3 hours incubation (i.e. photodynamic therapy (PDT)). Three settings are applied: mild, moderate and strong.
Drug: MAL Control. — Intervention: Topical application of 125 microliter methyl aminolevulinate (MAL) cream followed by red light illumination after 3 hours incubation (i.e. photodynamic therapy (PDT)).
Other: Untreated Control — Untreated control. No interventions.

SUMMARY:
The study investigates the potential of a range of different physical pretreatments to enhance methyl aminolevulinate (MAL)-induced protoporphyrin IX (PpIX) in the skin prior to photodynamic therapy (PDT).

DETAILED DESCRIPTION:
The study investigates the potential of a range of different physical pretreatments to enhance methyl aminolevulinate (MAL)-induced protoporphyrin IX (PpIX) in the skin prior to photodynamic therapy (PDT). The pretreatments include: microneedling, sandpaper, curettage, ablative fractional laser and non-ablative fractional laser. 17 treatment areas are mapped on the upper back of the participants. Each participant receives each intervention in a random sequence.

Primary outcome measure: PpIX accumulation after 3 hours incubation with MAL. Secondary outcome measures: pain during treatment and skin reactions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, healthy, fair skinned (skin type I-III)

Exclusion Criteria:

* Pregnant women
* Tattoos, moles or scars in treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Protoporphyrin IX (PpIX) fluorescence | Day 0
  Protoporphyrin IX (PpIX) fluorescence as measured by a fluorescence camera (Medeikonos PDD/PDT, Medeikonos AB,Gothenburg, Sweden).

SECONDARY OUTCOMES:
Pain | Day 0
  Pain during treatment as measured by Visual Analog Scale.
Skin reactions | Day 0, Day 1, Day 3, Day 7
  Skin reactions evaluated on a clinical scale.

REFERENCES:
- [Derived] Bay C, Lerche CM, Ferrick B, Philipsen PA, Togsverd-Bo K, Haedersdal M. Comparison of Physical Pretreatment Regimens to Enhance Protoporphyrin IX Uptake in Photodynamic Therapy: A Randomized Clinical Trial. JAMA Dermatol. 2017 Apr 1;153(4):270-278. doi: 10.1001/jamadermatol.2016.5268. PMID 28146245